CLINICAL TRIAL: NCT04340245
Title: Exploiting Risk-Based Risk Stratification in Early Prostate Cancer to Discriminate Progressors From Non-Progressors
Acronym: RECONCILE
Status: Active, not recruiting | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 127742
Record Dates: First submitted 2020-01-21; First posted 2020-04-09 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer
Keywords: MRI; MRI progression; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Sodium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, semen, prostate tissue from biopsy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: NA (Observational) — No interventions will be carried out. Comparisons will be made between patients whose cancer has progressed over the course of one year and patients whose cancer hasn't.

SUMMARY:
This study seeks to analyse MRI images and biological samples from 60 men diagnosed as having intermediate risk prostate cancer at baseline and one year afterwards to compare the molecular, genetic and transcriptomic differences between cancers that progress and cancers which do not.

DETAILED DESCRIPTION:
RECONCILE is a single centre, prospective, longitudinal observational cohort study. 60 consenting men with intermediate risk, gleason 3+4, prostate cancer under active surveillance will be recruited to the study. They will undergo blinded, concurrent molecular and radiological analysis of their cancer at baseline and at one year. Tests at baseline and one year will include mpMRI, targeted prostate biopsy and further tissue sampling (semen, urine and blood). There will be PSA monitoring at 3 monthly intervals throughout the study as per standard of care active surveillance. Tissue will be analysed for biological and molecular markers significantly associated with radiological progression events.

After consenting to taking part in the study a patient will come in for an MRI scan as standard of care. This scan will be used at a subsequent visit to inform a guided trans-perineal biopsy. At this biopsy visit patients will provide research blood samples, a urine sample and have a confirmatory biopsy. After the standard of care diagnostic tissue samples are taken, three research tissue samples will be taken.

If the patient has been identified through the ReIMAGINE study and consents to take part in RECONCILE then these baseline visits are not needed, the data from ReIMAGINE will be used as the baseline visit data.

The patient will come in as scheduled for their regular PSA visits in line with their active surveillance protocol. If a PSA test shows signs of potential progression the patient will have a standard of care diagnostic MRI, if this confirms progression then the imaging and biopsy visits scheduled for one year will be triggered early.

In the absence of any identified progression the patient will return after 12 months and have both the imaging and biopsy visits repeated (again providing blood and urine). After this visit the patient will be considered as having finished the study.

Patients who consent to take part in the study who have previously taken part in the PLiS semen donation study will be asked to provide a semen sample before the one year biopsy visit for comparison with the baseline sample that was provided for the PLiS study.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 18 years or above.
* Diagnosed with prostate cancer within 4 months of entry.
* Likert or PIRADS score greater than or equal to 4.
* PSA less than or equal to 15 ng.ml-1 in the last 6 months.
* mpMRI concordant with histology.
* Overall Gleason score 7 (3+4).
* Maximum cancer core length less than or equal to 10mm.
* Patients on active surveillance

Exclusion Criteria:

* Any contraindication to MRI scans (e.g. metal implants, unmanageable claustrophobia)
* Presence of a pacemaker
* Presence of a hip replacement
* Any hormonal treatment or inhibitors of 5 alpha-reductase in the previous 6 months
* Any previous TURP or other prostate surgery.
* Previous treatment for prostate cancer.
* Patients who have previously had sepsis due to a prostate biopsy
* Patients receiving concomitant treatment for their cancer
* Inability to provide full informed consent (e.g. due to dementia)

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must be men with prostate cancer
Study Population: Men over the age of 18 with prostate cancer (Gleason 3+4) who are on active surveillance.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion | 12 months
  Proportion of concordant pairs molecular progressor- radiological progressor.

SECONDARY OUTCOMES:
Progression time | 12 months
  Time to radiological progression
Lesion imaging characteristics | 12 months
  Quantitative and qualitative imaging characteristics of MRI lesions
Prostate imaging changes - quantitative | 12 months
  Quantitative imaging features (MRI and derivative) of MRI lesions(s), a radiological progression ring (if present) and the rest of the prostate at different time points
Prostate imaging changes - qualitative | 12 months
  Qualitative imaging features (MRI and derivative) of MRI lesion(s), a radiological progression ring (if present) and the rest of the prostate at different time points.
Imaging characteristics comparison | 12 months
  Quantitative imaging characteristics of MRI lesion(s), a radiological progression ring (if present) and the rest of the prostate at different time points and stratify by radiological progressors vs non progressors.
Histology | 12 months
  Qualitative and quantitative histologic composition of cancer and surrounding tissues
Heterogeneity | 12 months
  Histologic heterogeneity of cancer, both qualitatively and quantitatively
Molecular index | 12 months
  Molecular Index of cancer, peritumoral and normal tissue.
Urine and semen biomarkers | 12 months
  Next generation sequencing will be used to perform urinary and seminal genome, exosome, methylome and transcriptome analysis in order to identify novel molecular signatures associated with prostate cancer imaging endotypes. No commercial biomarkers will be assessed within this study.
  Biomarker definition (NIH NCI dictionary) A biological molecule found in blood, other body fluids, or tissues that is a sign of a normal or abnormal process, or of a condition or disease. A biomarker may be used to see how well the body responds to a treatment for a disease or condition. Also called molecular marker and signature molecule.
Inflammatory infiltrate | 12 months
  Qualitative and quantitative analysis of inflammatory infiltrate in cancer, peritumoral and normal tissue.
Blood biomarkers | 12 months
  Deep sequencing of circulating plasma DNA will be be used to explore novel prostate cancer biomarkers. Analysis of circulating inflammatory and immune markers including T-cell analysis will be used to correlate immunological biomarkers with prostate cancer endotypes.
Immune pathways | 12 months
  Qualitative and quantitative analysis of immune related pathways
Transition to active treatment | 12 months
  Proportion of patients who transition to active treatment, by time and type of treatment.
Treatment eligibility | 12 months
  Proportion of patients eligible to a type of treatment at baseline and follow-up.
Rate of metastasis | 12 months
  Rate of metastasis for prostate cancer at different time point.
Concordance, histology and imaging | 12 months
  Concordance rate between progression at histology and imaging.
Concordance, radiology | 12 months
  Concordance rate between radiologist for PRECISE scoring.
Patient reported outcomes - EPIC 26 | 12 months
  Patient reported outcomes at different time points using the RPIC 26 questionnaire
Patient reported outcomes - EORTC-QLQ-C30 | 12 months
  Patient reported outcomes at different time points using the EORTC-QLQ-C30 questionnaire
Patient reported outcomes - MAX-PC | 12 months
  Patient reported outcomes at different time points using the MAX-PC questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. Patients will be identified by a pseudo-anonymised patient number

REFERENCES:
- [Derived] Marsden T, Attard G, Punwani S, Giganti F, Freeman A, Haider A, Wingate A, Williams N, Syer T, Pashayan N, Moore CM, Emberton M, Orczyk C. The RECONCILE study protocol: Exploiting image-based risk stratification in early prostate cancer to discriminate progressors from non-progressors (RECONCILE). PLoS One. 2024 Oct 17;19(10):e0295994. doi: 10.1371/journal.pone.0295994. eCollection 2024. PMID 39418289